CLINICAL TRIAL: NCT05878327
Title: Livedoid Vasculopathy: Strong Association With Smoking, Weak Association With Thrombophilia
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH-Nr. 2013-0301
Record Dates: First submitted 2014-08-03; First posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Livedoid Vasculitis
Keywords: Livedoid Vasculitis; smoking; thrombophilia
MeSH Terms: conditions — Livedoid Vasculopathy; Smoking; Thrombophilia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood samples for thrombophilia screen.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Thrombophilia screening: Patients with livedoid vasculopathy. Investigated by thrombophilia screening
  Interventions: Other: Thrombophilia screening

INTERVENTIONS:
Other: Thrombophilia screening — No intervention. Blood is drawn for analysis.

SUMMARY:
A screening of patient histories at the clinics of Dermatology of the universities of Zurich, Basel and Bern is performed in order to identify patients with a history of Livedoid vasculopathy. Patients with a history of livedoid vasculopathy are asked to participate in the study. After reading the patient information and if the informed consent is signed patients are included in the study. Patients are questioned about their smoking history and blood is drawn in order to perform a screening for thrombophilia.

DETAILED DESCRIPTION:
A screening of patient histories at the clinics of Dermatology of the universities of Zurich, Basel and Bern is performed in order to identify patients with a history of Livedoid vasculopathy. Patients with a history of livedoid vasculopathy are asked to participate in the study. The presence of Livedoid vasculopathy must be confirmed by a histologic specimen. After reading the patient information and if the informed consent is signed patients are included in the study. Patients are questioned about their smoking history and blood is drawn in order to perform a screening for thrombophilia. The presence of a history of smoking and thrombophilia is compared to the general Swiss population.

ELIGIBILITY:
Inclusion Criteria:

* History of livedoid vasculopathy

Exclusion Criteria:

* Diagnosis was not proved by biopsy specimen
* A different reason than livedoid vasculopathy has been found for the symptoms of the patient
* No informed consent by the patient

Ages: 10 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated for livedoid vasculopathy at the clinics of Dermatology of the University hospitals of Zurich, Basel and Bern.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2013-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Smoking history: Patients will be asked if they currently smoke or if they are former smokers. If one of both items is yes, it means a positive answer. | 22 months
  The primary endpoint is the comparison of a positive smoking history and other cardiovascular risk factors of patients with livedoid vasculopathy with the Swiss general population.

SECONDARY OUTCOMES:
Thrombophilia screening: the following parameters will be determined in every participant: Factor V Leiden, Prothrombin 20210; Protein C, Protein S, Antithrombin III, Beta 2 Glykoprotein 1, Lupus Antikoagulans | 22 months
  The secondary endpoint is the search for thrombophilia in patients with livedoid vasculopathy.

CONTACTS AND LOCATIONS:
Overall Officials: Juerg Hafner, Prof, MD, Principal Investigator — University Hospital Zurich, Dept. of Dermatology
Locations (3):
- Switzerland (3):
  - University hospital of Basel, Basel
  - University hospital of Bern, Bern
  - University hospital Zurich, Zurich